CLINICAL TRIAL: NCT05164692
Title: Application of LiveSpo Navax in Treatment of Acute Respiratory Disease in Children Infected With Respiratory Syncytial Virus
Brief Title: Effects of Nasal-spraying LiveSpo Navax in Treatment of Acute Respiratory Infections in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Children's Hospital, Vietnam (Other)
Responsible Party: Principal Investigator, Tran Thanh Tu, Vice Director of International Center, Vietnam National Children's Hospital, National Children's Hospital, Vietnam
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020S-06; 4711/QD-BVNTU (Other: Vietnam National Children's Hospital)
Record Dates: First submitted 2021-12-06; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Acute Respiratory Tract Infections
Keywords: Respiratory Syncytial Virus (RSV); Acute Respiratory Tract Infections (ARTIs); Children; Nasal-spraying probiotics; Viral load; Co-infection bacteria; Cytokines; Bacillus spores

STUDY DESIGN:
Intervention Model Description: Blind, randomized, and controlled clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: LiveSpo Navax and placebo 0.9% NaCl physiological saline are indistinguishable regarding taste and smell. The color and turbidity of LiveSpo Navax suspension is unrecognizable to investigators except the PI and analyzer, nurses, patient's parents, and patients due to opaque plastic container.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Control group receives the routine treatment and uses 0.9% NaCl physiological saline:
  Routine treatment is as follows:
  * Oral administrative drugs: antipyretic paracetamol (Efferegant®️); anti-inflammatory corticosteroid methylprednisolon; antibiotics e.g. ampicillin and sulbactam complex (Ama-power®️), tobramycin (Medphatobra®️), or cefotaxim (Goldcefo®️), based on the results of antibiotic susceptibility test.
  * Aerosol therapy: bronchodilator e.g. salbutamol (Ventolin ®️inhaler) or budesonide (Pulmicort ®️Respules).
  Interventions: Drug: 0.9% NaCl physiological saline
- Navax (Experimental): Navax group receives the routine treatment and uses NaCl 0.9% plus B. subtilis and B. clausii at 5 billions CFU/5 mL (LiveSpo®️ Navax):
  Routine treatment is as follows:
  * Oral administrative drugs: antipyretic paracetamol (Efferegant®️); anti-inflammatory corticosteroid methylprednisolon; antibiotics e.g. ampicillin and sulbactam complex (Ama-power®️), tobramycin (Medphatobra®️), or cefotaxim (Goldcefo®️), based on the results of antibiotic susceptibility test.
  * Aerosol therapy: bronchodilator e.g. salbutamol (Ventolin ®️inhaler) or budesonide (Pulmicort ®️Respules).
  Interventions: Combination Product: LiveSpo Navax

INTERVENTIONS:
Combination Product: LiveSpo Navax — In Vietnam, LiveSpo Navax is manufactured as a Class-A medical device product (Product declaration No.210001337/PCBA-HN) under manufacturing standards approved by Hanoi Health Department, Ministry of Health, Vietnam (Certificate No YT117-19) and ISO 13485:2016.
  Other Names: Registration number: No.210001337/PCBA-HN
  Arms: Navax
Drug: 0.9% NaCl physiological saline — Nasal-spraying 0.9% NaCl physiological saline is prepared by extracting 5 mL from 0.9% NaCl intravenous infusion 500 mL PP bottle (B.Braun, Germany, product declaration No. VD-32732-19), and then pouring it into the same opaque plastic spraying 10 mL-bottle that is used for LiveSpo Navax.
  Other Names: Registration number: VD-32723-19
  Arms: Control

SUMMARY:
Rationals: Infection with the Respiratory Syncytial Virus (RSV) is one of the most common causes of respiratory tract diseases. However, treatment for pediatric RSV infection remains supportive to prevent co-infection bacteria and respiratory failure. In recent years, preventive and supportive probiotic therapies for respiratory tract infections (RTIs) have been increasingly strengthened, however, the use of oral administrative probiotics as functional foods is effective only for mild symptoms and not applicable for Acute RTIs (ARTIs). Here, we propose that direct spraying of probiotics into the nose can be a fast and effective symptomatic treatment for ARTIs.

Objectives: Investigate symptomatic treatment effects of probiotic product LiveSpo Navax, as liquid-suspension form containing Bacillus spores of safe B. subtilis ANA4 and B. clausii ANA39 strains, in children having acute respiratory diseases caused by RSV:

* Primary Objective: Evaluation of improved efficacy and reduced treatment time of LiveSpo Navax in children infected with RSV.
* Secondary Objectives: Measurement of changes in RSV viral load, co-infectious bacterial concentrations, and major cytokine indicators in the nasopharyngeal mucosa before and after 3 days using LiveSpo Navax.

Endpoints:

Primary endpoint: LiveSpo Navax alleviates RSV-infection symptoms about 25% more effectively, as indicated by 90% of patients using LiveSpo Navax (Navax group) are symptom-free at day 3-6 of intervention depending on symptoms, compared to 65% of patients in Control group.

Secondary endpoint: Patients in Navax group had more significant reductions in RSV load (>10 fold) than patients in Control group at day 3 of intervention.

Study Population: Sample size is 100. Description of Sites: The study is carried out at Vietnam National Children's Hospital.

Description of Study Intervention: Totally 100 eligible patients are divided randomly into 2 groups (n = 50/group each): Patients in Control group received the routine treatment and three times per day 0.9% NaCl physiological saline while the and patients in Navax group received three times per day LiveSpo Navax in addition to the same standard of care treatment. The standard treatment regimen is 3-6 days but can be extended further depending on the severity of the patients' respiratory failure.

Study Duration: 12 months

DETAILED DESCRIPTION:
Respiratory syncytial virus (RSV) is the most common virus that causes Acute Respiratory Tract Infections (ARTIs) in young children, with a high risk of serious bronchiolitis. RSV infection symptoms range from mild fever, cough, runny nose, and wheezing to severe symptoms such as difficulty breathing and respiratory failure. Cytokines in the airways of children with bronchiolitis, such as tumor necrosis factor (TNF-alpha), Interleukin-6 (IL-6) and IL-8, have been shown to increase at a very high level in primary RSV infection, and extreme elevation of IL-6 is associated with sudden death in children with RSV infection. The World Health Organization (WHO) estimates that 160,000-600,000 children under the age of five die or hospitalize each year as a result of RSV infection. There is currently no vaccine or specific treatment for RSV-infected children because monoclonal antibody palivizumab therapy and antiviral nucleotide drug ribavirin are either too expensive or too dangerous for children and are only recommended for high-risk patients.

In recent years, preventive and supportive therapies for respiratory tract infection have grown in popularity, with probiotics emerging as promising safe candidates for therapeutic support and antibiotic reduction. It is suggested that probiotics can capture viruses through direct interactions, or produce secondary growths that inhibit virus growth or stimulate the immune system to capture virus intrusion. However, the efficacy of oral digested probiotics on children's respiratory tracts has been slow to develop (normally it takes about 3-12 months) and is primarily used for prevention rather than supportive treatment of ARITs. As a result, alternative delivery routes for probiotics in the treatment of ARTIs are required.

The aim of the study about to evaluate the effectiveness of nasal-spraying probiotics containing two bacterial strains, Bacillus subtilis and Bacillus clausii in preventing and in supporting the treatment of children having acute respiratory symptoms due to RSV infection.

Methods: A randomized, blind, and controlled clinical trial are conducted. The patient's parents are required to provide the following information of their children: full name, sex, age, obstetric history, vaccination history, antibiotic use history… After informed consent, 100 patients with ARTIs due to RSV will be randomized into 2 groups (n = 50/group): the control group (named "Control" group) use 0.9% NaCl physiological saline and an experimental group (named the "Navax" group) use the probiotics LiveSpo Navax. The patient is given a coded spray in the form of a blind sample to ensure the objectivity of the study. The clinical follow-up will be 6 days, nasopharyngeal samples will be collected at day 0 and day 3 to evaluate potential reductions in viral load and co-infection bacteria, as well as modulation of overreacted cytokine release and the presence of probiotic spores in the patient's nasal mucosa.

Real-time PCR for detection of microorganism in nasopharyngeal samples: semi-quantitative assays for measuring changes in RSV load and co-infection bacterial concentrations is conducted by the real-time RT-PCR/PCR routine protocol which has been standardized under ISO 15189:2012 criteria and used in Vietnam National Children's Hospital. Detection of B. subtilis ANA4 and B. clausii ANA39 are also conducted by real-time PCR SYBR Green that has been standardized under ISO 17025: 2017 standard and routinely in the Key Laboratory of Enzyme and Protein Technology, VNU University of Science.

ELISA assays for cytokine levels: pro-inflammatory cytokines levels (pg/mL) including interleukin (IL-6, IL-8) and TNF-alpha are quantified using an enzyme-linked immunosorbent assay kit (ELISA) according to the manufacturer's instructions.

During treatment, patients are monitored daily for typical clinical symptoms of RSV-induced respiratory tract infections, including runny nose, chest depression, difficulty breathing, dry rales, moist rales, body temperature (oC), oxymetry (SpO2) (%), pulse (beats/min), and breath (beats/min) until discharged. The patients' health conditions are observed by doctors and nurses, and their pieces of information are filled in medical records. During this study, parents' patients are asked to abstain from consumption for their children of other probiotics, either via nasal spray or oral administration and refrain from cleaning nose for their children with other 0.9% NaCl physiological saline sprayers.

Data collection and statistical analysis: individual medical records are collected, and the patient's information is then gathered and systematized in a data set. The efficacy of LiveSpo Navax is evaluated and compared to 0.9% NaCl physiological saline based on the following clinical and sub-clinical criteria obtained in Navax and Control groups: (i) the symptomatic-relieving day; (ii) the reduction levels (2^△Ct) of RSV load and co-infection bacteria concentrations. △Ct for target genes is calculated as Ct (threshold cycle) at day 3 - Ct at day 0 while Ct of internal control is adjusted to be equal among all samples; (iii) the reduction levels of IL-6, IL-8, and TNF-alpha cytokines. The tabular analysis is performed on dichotomous variables using the χ2 test or Fisher's exact test when the expected value of any cell is below five. Continuous variables are compared using either the Wilcoxon test, t-test, or the Mann-Whitney test when data are not normally distributed. The correlations among the variables are assessed by Spearman's correlation analysis. Statistical and graphical analyses are performed on GraphPad Prism v8.4.3 software (GraphPad Software, CA, USA). The significance level of all analyzes is set at p < 0.05. P-values.

Expected outcomes: (i) LiveSpo Navax alleviates RSV-infection symptoms about 25% more effectively, as indicated by 90% of patients using LiveSpo Navax (Navax group) are symptom-free at day 3-6 of intervention depending on symptoms, compared to 65% of patients in Control group; (ii) Patients in Navax group has more significant reductions in RSV load (>10 fold) than patients in Control group at day 3 of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Children (male/female) aged from 4 to 60 months.
* Admitted hospital due to lower respiratory infection.
* RSV is positive by rapid test.
* Parents of the pediatric patient agree to participate in the study, explain and sign the research consent form.

Exclusion Criteria:

* Newborn babies.
* Have a history of drug allergy.
* Need oxygen therapy.
* Discharged before day 3.
* Lost to follow-up.
* Withdrawn from the trial.
* Continuing in the trial but missing data.
* Meeting the criteria for psychiatric disorders other than depression and/or anxiety.

Ages: 4 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2020-08-29 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2021-08-29 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with free respiratory symptoms | Day 0 to day 6
  Percentage (%) of RSV-infected patients with free respiratory symptoms including runny nose, chest depression, difficulty breathing, dry rales, and moist rales

SECONDARY OUTCOMES:
Patient's breath | Day 0 to day 6
  RSV-infected patient's breath (beats/min) before and after nasal-spraying
Patient's pulse | Day 0 to day 6
  RSV-infected patient's pulse (beats/min) before and after nasal-spraying
Patient's temperature | Day 0 to day 6
  RSV-infected patient's temperature (oC) before and after nasal-spraying
Patient's pulse oxygen (SpO2) | Day 0 to day 6
  RSV-infected patient's pulse oxygen-SpO2 (%) before and after nasal-spraying
RSV concentration | Day 0 and day 3
  Concentration of respiratory syncytial virus in nasopharyngeal samples, as indicated by real time PCR threshold cycle (Ct) value
Co-infection bacterial concentrations | Day 0 and day 3
  Co-infection bacterial concentrations in nasopharyngeal samples, as indicated by real time PCR threshold cycle (Ct) values
Cytokines levels | Day 0 and day 3
  Levels (pg/mL) of tumor necrosis factor-α (TNF-α), interleukin-6 (IL-6), and interleukin-8 (IL-8) in nasopharyngeal samples

CONTACTS AND LOCATIONS:
Overall Officials: Tu T Tran, PhD. MD., Principal Investigator — International Center, Vietnam National Children's Hospital
Locations (1):
- International Center, Vietnam National Children's Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Data or samples share that will be coded, with no PHI include. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research and will be provided following review and approval of a study protocol, informed consent form (ICF), clinical study peport (CSR). For more information or to submit a request, please contact clinicaltrial.probiotics@gmail.com

REFERENCES:
- [Result] Lima SF, Teixeira AG, Higgins CH, Lima FS, Bicalho RC. The upper respiratory tract microbiome and its potential role in bovine respiratory disease and otitis media. Sci Rep. 2016 Jul 1;6:29050. doi: 10.1038/srep29050. PMID 27363739
- [Result] Chotirmall SH, Gellatly SL, Budden KF, Mac Aogain M, Shukla SD, Wood DL, Hugenholtz P, Pethe K, Hansbro PM. Microbiomes in respiratory health and disease: An Asia-Pacific perspective. Respirology. 2017 Feb;22(2):240-250. doi: 10.1111/resp.12971. PMID 28102970
- [Result] Principi N, Cozzali R, Farinelli E, Brusaferro A, Esposito S. Gut dysbiosis and irritable bowel syndrome: The potential role of probiotics. J Infect. 2018 Feb;76(2):111-120. doi: 10.1016/j.jinf.2017.12.013. Epub 2017 Dec 29. PMID 29291933
- [Result] Sonawane AR, Tian L, Chu CY, Qiu X, Wang L, Holden-Wiltse J, Grier A, Gill SR, Caserta MT, Falsey AR, Topham DJ, Walsh EE, Mariani TJ, Weiss ST, Silverman EK, Glass K, Liu YY. Microbiome-Transcriptome Interactions Related to Severity of Respiratory Syncytial Virus Infection. Sci Rep. 2019 Sep 25;9(1):13824. doi: 10.1038/s41598-019-50217-w. PMID 31554845
- [Result] Li KJ, Chen ZL, Huang Y, Zhang R, Luan XQ, Lei TT, Chen L. Dysbiosis of lower respiratory tract microbiome are associated with inflammation and microbial function variety. Respir Res. 2019 Dec 3;20(1):272. doi: 10.1186/s12931-019-1246-0. PMID 31796027
- [Result] Valdivieso-Ugarte M, Gomez-Llorente C, Plaza-Diaz J, Gil A. Antimicrobial, Antioxidant, and Immunomodulatory Properties of Essential Oils: A Systematic Review. Nutrients. 2019 Nov 15;11(11):2786. doi: 10.3390/nu11112786. PMID 31731683
- [Result] Elshaghabee FMF, Rokana N, Gulhane RD, Sharma C, Panwar H. Bacillus As Potential Probiotics: Status, Concerns, and Future Perspectives. Front Microbiol. 2017 Aug 10;8:1490. doi: 10.3389/fmicb.2017.01490. eCollection 2017. PMID 28848511
- [Result] Raveendran S, Parameswaran B, Ummalyma SB, Abraham A, Mathew AK, Madhavan A, Rebello S, Pandey A. Applications of Microbial Enzymes in Food Industry. Food Technol Biotechnol. 2018 Mar;56(1):16-30. doi: 10.17113/ftb.56.01.18.5491. PMID 29795993
- [Result] Yang L, Zeng X, Qiao S. Advances in research on solid-state fermented feed and its utilization: The pioneer of private customization for intestinal microorganisms. Anim Nutr. 2021 Dec;7(4):905-916. doi: 10.1016/j.aninu.2021.06.002. Epub 2021 Sep 16. PMID 34632121
- [Result] Oggioni MR, Pozzi G, Valensin PE, Galieni P, Bigazzi C. Recurrent septicemia in an immunocompromised patient due to probiotic strains of Bacillus subtilis. J Clin Microbiol. 1998 Jan;36(1):325-6. doi: 10.1128/JCM.36.1.325-326.1998. No abstract available. PMID 9431982
- [Result] Cukovic-Cavka S, Likic R, Francetic I, Rustemovic N, Opacic M, Vucelic B. Lactobacillus acidophilus as a cause of liver abscess in a NOD2/CARD15-positive patient with Crohn's disease. Digestion. 2006;73(2-3):107-10. doi: 10.1159/000094041. Epub 2006 Jun 20. PMID 16788305
- [Result] Borriello SP, Hammes WP, Holzapfel W, Marteau P, Schrezenmeir J, Vaara M, Valtonen V. Safety of probiotics that contain lactobacilli or bifidobacteria. Clin Infect Dis. 2003 Mar 15;36(6):775-80. doi: 10.1086/368080. Epub 2003 Mar 5. PMID 12627362
- [Result] Song M, Hong HA, Huang JM, Colenutt C, Khang DD, Nguyen TV, Park SM, Shim BS, Song HH, Cheon IS, Jang JE, Choi JA, Choi YK, Stadler K, Cutting SM. Killed Bacillus subtilis spores as a mucosal adjuvant for an H5N1 vaccine. Vaccine. 2012 May 9;30(22):3266-77. doi: 10.1016/j.vaccine.2012.03.016. Epub 2012 Mar 22. PMID 22446640
- [Result] Hong JE, Kye YC, Park SM, Cheon IS, Chu H, Park BC, Park YM, Chang J, Cho JH, Song MK, Han SH, Yun CH. Alveolar Macrophages Treated With Bacillus subtilis Spore Protect Mice Infected With Respiratory Syncytial Virus A2. Front Microbiol. 2019 Mar 12;10:447. doi: 10.3389/fmicb.2019.00447. eCollection 2019. PMID 30930867
- [Result] Lefevre M, Racedo SM, Ripert G, Housez B, Cazaubiel M, Maudet C, Justen P, Marteau P, Urdaci MC. Probiotic strain Bacillus subtilis CU1 stimulates immune system of elderly during common infectious disease period: a randomized, double-blind placebo-controlled study. Immun Ageing. 2015 Dec 3;12:24. doi: 10.1186/s12979-015-0051-y. eCollection 2015. PMID 26640504
- [Result] Tavares Batista M, Souza RD, Paccez JD, Luiz WB, Ferreira EL, Cavalcante RC, Ferreira RC, Ferreira LC. Gut adhesive Bacillus subtilis spores as a platform for mucosal delivery of antigens. Infect Immun. 2014 Apr;82(4):1414-23. doi: 10.1128/IAI.01255-13. Epub 2014 Jan 13. PMID 24421038
- [Result] Fazle Rabbee M, Baek KH. Antimicrobial Activities of Lipopeptides and Polyketides of Bacillus velezensis for Agricultural Applications. Molecules. 2020 Oct 27;25(21):4973. doi: 10.3390/molecules25214973. PMID 33121115
- [Result] Marseglia GL, Tosca M, Cirillo I, Licari A, Leone M, Marseglia A, Castellazzi AM, Ciprandi G. Efficacy of Bacillus clausii spores in the prevention of recurrent respiratory infections in children: a pilot study. Ther Clin Risk Manag. 2007 Mar;3(1):13-7. doi: 10.2147/tcrm.2007.3.1.13. PMID 18360611
- [Result] Piewngam P, Zheng Y, Nguyen TH, Dickey SW, Joo HS, Villaruz AE, Glose KA, Fisher EL, Hunt RL, Li B, Chiou J, Pharkjaksu S, Khongthong S, Cheung GYC, Kiratisin P, Otto M. Pathogen elimination by probiotic Bacillus via signalling interference. Nature. 2018 Oct;562(7728):532-537. doi: 10.1038/s41586-018-0616-y. Epub 2018 Oct 10. PMID 30305736
- [Result] Collins PL, Murphy BR. Respiratory syncytial virus: reverse genetics and vaccine strategies. Virology. 2002 May 10;296(2):204-11. doi: 10.1006/viro.2002.1437. No abstract available. PMID 12069519
- [Result] Nguyen SN, Nguyen TNT, Vu LT, Nguyen TD. Clinical Epidemiological Characteristics and Risk Factors for Severe Bronchiolitis Caused by Respiratory Syncytial Virus in Vietnamese Children. Int J Pediatr. 2021 Nov 15;2021:9704666. doi: 10.1155/2021/9704666. eCollection 2021. PMID 34819958
- [Result] Wang X, Li Y, Deloria-Knoll M, Madhi SA, Cohen C, Ali A, Basnet S, Bassat Q, Brooks WA, Chittaganpitch M, Echavarria M, Fasce RA, Goswami D, Hirve S, Homaira N, Howie SRC, Kotloff KL, Khuri-Bulos N, Krishnan A, Lucero MG, Lupisan S, Mira-Iglesias A, Moore DP, Moraleda C, Nunes M, Oshitani H, Owor BE, Polack FP, O'Brien KL, Rasmussen ZA, Rath BA, Salimi V, Scott JAG, Simoes EAF, Strand TA, Thea DM, Treurnicht FK, Vaccari LC, Yoshida LM, Zar HJ, Campbell H, Nair H; Respiratory Virus Global Epidemiology Network. Global burden of acute lower respiratory infection associated with human metapneumovirus in children under 5 years in 2018: a systematic review and modelling study. Lancet Glob Health. 2021 Jan;9(1):e33-e43. doi: 10.1016/S2214-109X(20)30393-4. Epub 2020 Nov 26. PMID 33248481
- [Result] Griffiths C, Drews SJ, Marchant DJ. Respiratory Syncytial Virus: Infection, Detection, and New Options for Prevention and Treatment. Clin Microbiol Rev. 2017 Jan;30(1):277-319. doi: 10.1128/CMR.00010-16. PMID 27903593
- [Result] Kakimoto Y, Seto Y, Ochiai E, Satoh F, Osawa M. Cytokine Elevation in Sudden Death With Respiratory Syncytial Virus: A Case Report of 2 Children. Pediatrics. 2016 Dec;138(6):e20161293. doi: 10.1542/peds.2016-1293. Epub 2016 Nov 10. PMID 27940684
- [Result] Caly L, Ghildyal R, Jans DA. Respiratory virus modulation of host nucleocytoplasmic transport; target for therapeutic intervention? Front Microbiol. 2015 Aug 14;6:848. doi: 10.3389/fmicb.2015.00848. eCollection 2015. PMID 26322040
- [Result] Shi T, McAllister DA, O'Brien KL, Simoes EAF, Madhi SA, Gessner BD, Polack FP, Balsells E, Acacio S, Aguayo C, Alassani I, Ali A, Antonio M, Awasthi S, Awori JO, Azziz-Baumgartner E, Baggett HC, Baillie VL, Balmaseda A, Barahona A, Basnet S, Bassat Q, Basualdo W, Bigogo G, Bont L, Breiman RF, Brooks WA, Broor S, Bruce N, Bruden D, Buchy P, Campbell S, Carosone-Link P, Chadha M, Chipeta J, Chou M, Clara W, Cohen C, de Cuellar E, Dang DA, Dash-Yandag B, Deloria-Knoll M, Dherani M, Eap T, Ebruke BE, Echavarria M, de Freitas Lazaro Emediato CC, Fasce RA, Feikin DR, Feng L, Gentile A, Gordon A, Goswami D, Goyet S, Groome M, Halasa N, Hirve S, Homaira N, Howie SRC, Jara J, Jroundi I, Kartasasmita CB, Khuri-Bulos N, Kotloff KL, Krishnan A, Libster R, Lopez O, Lucero MG, Lucion F, Lupisan SP, Marcone DN, McCracken JP, Mejia M, Moisi JC, Montgomery JM, Moore DP, Moraleda C, Moyes J, Munywoki P, Mutyara K, Nicol MP, Nokes DJ, Nymadawa P, da Costa Oliveira MT, Oshitani H, Pandey N, Paranhos-Baccala G, Phillips LN, Picot VS, Rahman M, Rakoto-Andrianarivelo M, Rasmussen ZA, Rath BA, Robinson A, Romero C, Russomando G, Salimi V, Sawatwong P, Scheltema N, Schweiger B, Scott JAG, Seidenberg P, Shen K, Singleton R, Sotomayor V, Strand TA, Sutanto A, Sylla M, Tapia MD, Thamthitiwat S, Thomas ED, Tokarz R, Turner C, Venter M, Waicharoen S, Wang J, Watthanaworawit W, Yoshida LM, Yu H, Zar HJ, Campbell H, Nair H; RSV Global Epidemiology Network. Global, regional, and national disease burden estimates of acute lower respiratory infections due to respiratory syncytial virus in young children in 2015: a systematic review and modelling study. Lancet. 2017 Sep 2;390(10098):946-958. doi: 10.1016/S0140-6736(17)30938-8. Epub 2017 Jul 7. PMID 28689664
- [Result] Shahbazi R, Yasavoli-Sharahi H, Alsadi N, Ismail N, Matar C. Probiotics in Treatment of Viral Respiratory Infections and Neuroinflammatory Disorders. Molecules. 2020 Oct 22;25(21):4891. doi: 10.3390/molecules25214891. PMID 33105830
- [Result] Lehtoranta L, Pitkaranta A, Korpela R. Probiotics in respiratory virus infections. Eur J Clin Microbiol Infect Dis. 2014 Aug;33(8):1289-302. doi: 10.1007/s10096-014-2086-y. Epub 2014 Mar 18. PMID 24638909
- [Result] Starosila D, Rybalko S, Varbanetz L, Ivanskaya N, Sorokulova I. Anti-influenza Activity of a Bacillus subtilis Probiotic Strain. Antimicrob Agents Chemother. 2017 Jun 27;61(7):e00539-17. doi: 10.1128/AAC.00539-17. Print 2017 Jul. PMID 28416546
- [Result] Salminen S, Collado MC, Endo A, Hill C, Lebeer S, Quigley EMM, Sanders ME, Shamir R, Swann JR, Szajewska H, Vinderola G. The International Scientific Association of Probiotics and Prebiotics (ISAPP) consensus statement on the definition and scope of postbiotics. Nat Rev Gastroenterol Hepatol. 2021 Sep;18(9):649-667. doi: 10.1038/s41575-021-00440-6. Epub 2021 May 4. PMID 33948025
- [Result] Anderson LJ, Dormitzer PR, Nokes DJ, Rappuoli R, Roca A, Graham BS. Strategic priorities for respiratory syncytial virus (RSV) vaccine development. Vaccine. 2013 Apr 18;31 Suppl 2(Suppl 2):B209-15. doi: 10.1016/j.vaccine.2012.11.106. PMID 23598484
- [Result] Domachowske JB, Anderson EJ, Goldstein M. The Future of Respiratory Syncytial Virus Disease Prevention and Treatment. Infect Dis Ther. 2021 Mar;10(Suppl 1):47-60. doi: 10.1007/s40121-020-00383-6. Epub 2021 Mar 3. PMID 33656652
- [Result] Arnold R, Humbert B, Werchau H, Gallati H, Konig W. Interleukin-8, interleukin-6, and soluble tumour necrosis factor receptor type I release from a human pulmonary epithelial cell line (A549) exposed to respiratory syncytial virus. Immunology. 1994 May;82(1):126-33. PMID 7519169
- [Result] Ugonna K, Douros K, Bingle CD, Everard ML. Cytokine responses in primary and secondary respiratory syncytial virus infections. Pediatr Res. 2016 Jun;79(6):946-50. doi: 10.1038/pr.2016.29. Epub 2016 Feb 16. PMID 26882371
- See also: Novel insight on probiotic Bacillus subtilis: mechanism of action and clinical applications. — https://doi.org/10.4103/2455-3069.198381